CLINICAL TRIAL: NCT04041765
Title: Efficacy of Prophylactic IgM-Enriched Immunoglobulin for the Management of Early-Onset Neonatal Sepsis in Very Low Birth Weight Preterm Neonates; A Randomized Controlled Trial
Brief Title: IgM-Enriched Immunoglobulin for Neonatal Sepsis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fakultas Kedokteran Universitas Indonesia (Other)
Responsible Party: Principal Investigator, Rinawati, Principal Investigator; Senior Clinical Staff of Perinatology Division, Department of Child Health, Cipto Mangunkusumo Hospital; Head of Kiara Center of Maternal and Child Health, Cipto Mangunkusumo Hospital, Fakultas Kedokteran Universitas Indonesia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 19-11-432
Record Dates: First submitted 2019-07-27; First posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Neonatal Sepsis, Early-Onset; Very Low Birth Weight Infant; Inflammation; Infant, Newborn, Disease
Keywords: IgM-enriched Intravenous Immunoglobulin
MeSH Terms: conditions — Neonatal Sepsis; Inflammation; Disease | interventions — pentaglobulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): IgM-enriched IVIG given with dose of 0.25g/kg over 3 hours for 3 days in addition to Antibiotics
  Interventions: Drug: IgM-enriched IVIG
- Placebo Group (Placebo Comparator): Antibiotics only
  Interventions: Drug: IgM-enriched IVIG

INTERVENTIONS:
Drug: IgM-enriched IVIG — Contains human plasma protein 50mg/ml. With composition of Immunoglobulin M (IgM) 6mg, Immunoglobulin A (IgA) 6mg, Immunoglobulin G (IgG) 38mg (IgG subcl. approx. 63 % IgG1, 26 % IgG2, 4 % IgG3 and 7 % IgG4), Glucose monohydrate, sodium chloride, water for injections
  Other Names: Pentaglobin®

SUMMARY:
This study compares giving prophylactic IgM enriched Intravenous Immunoglobulin (IVIG) with placebo in 1 hour after birth, in neonates with risk factors of Early-Onset Neonatal Sepsis (EONS). In addition to the intervention, standard regimen antibiotics are also given within 1 hour. The IVIG is given for 3 days and primary and secondary outcomes will be collected. Risk factors are both from maternal and neonate origin.

DETAILED DESCRIPTION:
This randomized-controlled trial conducted in Cipto Mangunkusumo Hospital, Jakarta, Indonesia aims to determine the efficacy of prophylactic IgM-Enriched IVIG in preventing EONS. A total of 70 very low birth weight (VLBW) neonates with risk factors for EONS including maternal factors of premature rupture of membrane (PROM), fever, urinary tract infection (UTI), chorioamnionitis, and neonatal factor of prematurity and resuscitation history will be collected. These neonates within 1 hour of life will then be administered either placebo or IgM-enriched IVIG 0.25g/kg/day for 3 days, in addition to first-line empiric antibiotic. Randomization is done using simple randomization. Triple masking (Participant, Investigator, Outcomes Assessor) is conducted.

These neonates will then be clinically observed and evaluated for early mortality (mortality below 7 days), hemodynamics, length of stay, blood culture results, C-Reactive Protein (CRP), IT ratio, routine hematological examination, and IgGAME as parameters of improvement and prevention of EONS.

STATA version 12 (Macintosh version) will be used for data management and statistical analyses. The variables will first be presented descriptively, continued with bivariate and multivariate analysis. Bivariate analysis will be conducted between independent and dependent variables using chi-square/Fisher's exact test, Student's t-test, and Kruskal-Wallis. Variables with p-values <0.25 will be included in the multivariate analysis using logistic regression. The investigators will use two-sided p-values in our analysis with a p < 0.05 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants (< 1500 g)
* Gestational age below 32 weeks
* Risk of Early-Onset sepsis from maternal and neonate factors
* Inborn neonates

Exclusion Criteria:

* Birth weight < 600 g
* Gestational age < 26 weeks
* Multiple Congenital Anomaly
* Neonates with suspected congenital syndrome

Ages: 1 Minute to 1 Hour | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Early Mortality Rate | 1 week
  Neonates in the treatment group should have lower mortality rate in the first week of life

SECONDARY OUTCOMES:
Positive blood culture | 1 week
  Neonates in the treatment group should have less number of positive blood culture than those in the place group
Duration of NICU stay | Through study completion, an average of 3 months
  Neonates in the treatment group should be discharged earlier than those in the placebo group
Quantitative CRP Levels | 1 week
  Neonates in the treatment group should have lower CRP levels than those in the placebo group
IT Ratio value | 1 week
  Neonates in the treatment group should have lower IT Ratio value than those in the placebo group
Leukocyte count | 1 week
  Neonates in the treatment group should have lower Leukocyte count than those in the placebo group
IgGAME (IgG, IgM, IgA, IgE) Levels | 1 week
  Neonates in the treatment group should have higher IgGAME levels than those in the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Rinawati Rohsiswatmo, MD, PhD, Study Chair — Faculty of Medicine, Universitas Indonesia - Cipto Mangunkusumo Hospital; Nina D Putri, MD, PhD, Principal Investigator — Faculty of Medicine, Universitas Indonesia - Cipto Mangunkusumo Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capasso L, Borrelli AC, Parrella C, Lama S, Ferrara T, Coppola C, Catania MR, Iula VD, Raimondi F. Are IgM-enriched immunoglobulins an effective adjuvant in septic VLBW infants? Ital J Pediatr. 2013 Oct 7;39:63. doi: 10.1186/1824-7288-39-63. PMID 24098953
- [Background] Haque KN, Zaidi MH, Bahakim H. IgM-enriched intravenous immunoglobulin therapy in neonatal sepsis. Am J Dis Child. 1988 Dec;142(12):1293-6. doi: 10.1001/archpedi.1988.02150120047038. PMID 3195529
- [Background] Reith HB, Rauchschwalbe SK, Mittelkotter U, Engemann R, Thiede A, Arnold A, Lissner R. IgM-enriched immunoglobulin (pentaglobin) positively influences the course of post-surgical intra-abdominal infections. Eur J Med Res. 2004 Oct 29;9(10):479-84. PMID 15546815
- [Background] Capasso L, Borrelli AC, Pirozzi MR, Bucci L, Albachiara R, Ferrara T, Raimondi F. IgM and IgA enriched polyclonal immunoglobulins reduce short term mortality in extremely low birth weight infants with sepsis: a retrospective cohort study. Minerva Pediatr (Torino). 2021 Feb;73(1):3-7. doi: 10.23736/S2724-5276.18.04850-8. Epub 2018 Feb 19. PMID 29460549
- [Background] Capasso L, Borrelli AC, Ferrara T, Coppola C, Cerullo J, Izzo F, Caiazza R, Lama S, Raimondi F. Immunoglobulins in neonatal sepsis: has the final word been said? Early Hum Dev. 2014 Sep;90 Suppl 2:S47-9. doi: 10.1016/S0378-3782(14)50013-8. PMID 25220128